CLINICAL TRIAL: NCT00006359
Title: Phase II Trial of Androgen Suppression for 6 Months Combined With External Beam Radiotherapy (EBRT) With Brachytherapy (BT) Boost for Intermediate Risk Prostate Cancer
Brief Title: Androgen Suppression Plus Radiation Therapy in Treating Patients With Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CALGB-99809; U10CA031946 (NIH); CALGB-99809; CDR0000068228 (Registry Identifier: NCI Physician Data Query)
Record Dates: First submitted 2000-10-04; First posted 2003-01-27 (Estimated); Last update posted 2016-07-18 (Estimated); Status verified 2016-07

CONDITIONS: Prostate Cancer
Keywords: adenocarcinoma of the prostate; stage I prostate cancer; stage II prostate cancer; stage III prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Gonadotropin-Releasing Hormone; Androgen Antagonists; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Androgen suppression + EBRT + Brachytherapy (Experimental): Androgen suppression with external beam radiation therapy followed by brachytherapy boost
  Interventions: Drug: LHRH agonist; Drug: antiandrogen; Radiation: radiation therapy; Radiation: Brachytherapy boost

INTERVENTIONS:
Drug: LHRH agonist — Lupron: 22.5mg IM injection q 12 wks x 2 OR Zoladex: 10.8 mg subQ injection q 12 wks x 2
Drug: antiandrogen — flutamide 250 mg PO tid for 4 wks OR casodex 50 mg PO daily for 4 wks
Radiation: radiation therapy — 4500 cGy total dose given days 1-5 for 5 weeks following initiation of androgen suppression (25 fractions)
Radiation: Brachytherapy boost — Iodine 125 0.3 to 0.5 U per seed OR palladium 103 1.04 to 1.4 U per seed as implant; prescribed dose of I-125 100 Gy (TG-43) and Pd-103 90 Gy

SUMMARY:
RATIONALE: Androgens can cause the growth of prostate cancer cells. Drugs, such as leuprolide, goserelin, flutamide, or bicalutamide, may stop the adrenal glands from making androgens. Radiation therapy uses high-energy x-rays to damage tumor cells. Giving these drugs together with radiation therapy may kill more tumor cells.

PURPOSE: This phase II trial is studying how well androgen suppression with either leuprolide or goserelin and either flutamide or bicalutamide together with radiation therapy works in treating patients with prostate cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the feasibility of androgen-suppression therapy combined with external-beam radiotherapy and boost brachytherapy (EBRT+BT) in patients with intermediate-risk localized prostate cancer.
* Determine the safety of EBRT+BT in these patients.
* Determine, in a preliminary manner, the efficacy of EBRT+BT in terms of rate of local recurrence at 5 years, time to prostate-specific antigen failure, and time to first rectal/bladder injury, in these patients.

OUTLINE: Patients receive either leuprolide intramuscularly or goserelin subcutaneously once every 12 weeks for a total of 24 weeks. Patients also receive either oral flutamide three times daily or oral bicalutamide once daily for 4 weeks.

Within 4 weeks after initiation of androgen-suppression therapy, patients undergo external-beam radiotherapy (EBRT) once daily, 5 days a week, for 5 weeks. At 2-4 weeks after completion of EBRT, patients undergo transrectal ultrasound-guided boost brachytherapy with implanted iodine I 125 or palladium Pd 103 seeds.

Patients are followed every 3 months for 2 years and then every 6 months for 4 years.

PROJECTED ACCRUAL: A total of 60 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed adenocarcinoma of the prostate

  * Must have one of the following prognostic factors:

    * Stage T1-2, N0; prostate-specific antigen (PSA) ≤ 10 ng/mL; and Gleason score > 6
    * Stage T1-2, N0; PSA > 10 ng/mL and < 20 ng/mL; and Gleason score ≤ 6
    * Stage T3a, N0; PSA ≤ 10 ng/mL; and Gleason score ≤ 6
* Prostate volume < 60 cc by transrectal ultrasound
* No distant or nodal metastases

  * No metastatic disease by bone scan, CT scan, or MRI

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* ECOG 0-2

Life expectancy:

* Not specified

Hematopoietic:

* Absolute neutrophil count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3

Hepatic:

* Bilirubin ≤ 1.5 times upper limit of normal

Renal:

* Not specified

Other:

* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* No prior immunotherapy for prostate cancer

Chemotherapy:

* No prior chemotherapy for prostate cancer

Endocrine therapy:

* Prior androgen-suppression therapy for up to 4 weeks duration allowed if initiated within 4 weeks of study radiotherapy
* No other prior hormonal therapy

Radiotherapy:

* No prior radiotherapy for prostate cancer

Surgery:

* No prior surgery for prostate cancer
* No prior transurethral resection of the prostate

Other:

* No prior alternative therapy (e.g., PC-SPES) for prostate cancer

Ages: 18 Years to 120 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2000-09; Primary Completion 2007-10 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Toxicity | q 3 mon for 2 yrs post tx initiation

SECONDARY OUTCOMES:
Time to PSA failure | 6 years
Survival | 6 years
  Progression free and overall survival will be assessed

CONTACTS AND LOCATIONS:
Overall Officials: Mark Hurwitz, MD, Study Chair — Dana-Farber/Brigham and Women's Cancer Center
Locations (26):
- United States (26):
  - Beebe Medical Center, Lewes, Delaware
  - CCOP - Christiana Care Health Services, Newark, Delaware
  - St. Francis Hospital, Wilmington, Delaware
  - Florida Hospital Cancer Institute at Florida Hospital Orlando, Orlando, Florida
  - Union Hospital Cancer Center at Union Hospital, Elkton MD, Maryland
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Dana-Farber/Harvard Cancer Center at Dana Farber Cancer Institute, Boston, Massachusetts
  - Hudner Oncology Center at Saint Anne's Hospital, Fall River, Massachusetts
  - UMASS Memorial Cancer Center - University Campus, Worcester, Massachusetts
  - Ellis Fischel Cancer Center at University of Missouri - Columbia, Columbia, Missouri
  - CCOP - Kansas City, Kansas City, Missouri
  - Missouri Baptist Cancer Center, St Louis, Missouri
  - Arch Medical Services, Incoroporated at Center for Cancer Care Research, St Louis, Missouri
  - Washoe Cancer Services at Washoe Medical Center - Reno, Reno, Nevada
  - Cancer Institute of New Jersey at the Cooper University Hospital - Voorhees, Camden, New Jersey
  - Roswell Park Cancer Institute, Buffalo, New York
  - CCOP - Syracuse Hematology-Oncology Associates of Central New York, P.C., Syracuse, New York
  - SUNY Upstate Medical University Hospital, Syracuse, New York
  - Veterans Affairs Medical Center - Syracuse, Syracuse, New York
  - Community General Hospital of Greater Syracuse, Syracuse, New York
  - Presbyterian Cancer Center at Presbyterian Hospital, Charlotte, North Carolina
  - Wayne Memorial Hospital, Incorporated, Goldsboro, North Carolina
  - Zimmer Cancer Center at New Hanover Regional Medical Center, Wilmington, North Carolina
  - Comprehensive Cancer Center at Wake Forest University, Winston-Salem, North Carolina
  - Arthur G. James Cancer Hospital and Solove Research Institute at Ohio State University, Columbus, Ohio
  - Danville Regional Medical Center, Danville, Virginia

REFERENCES:
- [Result] Hurwitz MD, Halabi S, Archer L, et al.: Combination external beam radiation and brachytherapy boost with androgen suppression for treatment of intermediate-risk prostate cancer: long-term results of CALGB 99809. [Abstract] 2010 Genitourinary Cancers Symposium, March 5-7, 2010, San Francisco, California. A-192, 2010.
- [Result] Hurwitz MD, Halabi S, Ou SS, McGinnis LS, Keuttel MR, Dibiase SJ, Small EJ. Combination external beam radiation and brachytherapy boost with androgen suppression for treatment of intermediate-risk prostate cancer: an initial report of CALGB 99809. Int J Radiat Oncol Biol Phys. 2008 Nov 1;72(3):814-9. doi: 10.1016/j.ijrobp.2008.01.010. Epub 2008 Apr 11. PMID 18407435